CLINICAL TRIAL: NCT02467621
Title: Stress Ulcer Prophylaxis in the Intensive Care Unit (SUP-ICU)
Brief Title: Stress Ulcer Prophylaxis in the Intensive Care Unit
Acronym: SUP-ICU
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Dr. Morten Hylander Møller (Other)
Collaborators: Rigshospitalet, Denmark (Other); Copenhagen Trial Unit, Center for Clinical Intervention Research (Other)
Responsible Party: Sponsor-Investigator, Dr. Morten Hylander Møller, Principal investigator, Scandinavian Critical Care Trials Group
Organization: Scandinavian Critical Care Trials Group (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: RH-ITA-006
Record Dates: First submitted 2015-06-05; First posted 2015-06-10 (Estimated); Results first posted 2019-06-07 (Actual); Last update posted 2022-11-15 (Actual); Status verified 2022-10

CONDITIONS: Gastrointestinal Bleeding; Stress Ulcers
Keywords: Stress ulcer prophylaxis; Proton pump inhibitor; Pneumonia; Clostridium difficile infection
MeSH Terms: conditions — Gastrointestinal Hemorrhage; Duodenal Ulcer; Pneumonia; Clostridium Infections | interventions — Pantoprazole; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Proton pump inhibitor (PPI) (Experimental): Pantoprazole 40 mg
  Interventions: Drug: Pantoprazole
- Normal saline (Placebo Comparator): Saline (0.9%)
  Interventions: Other: Saline (0.9%)

INTERVENTIONS:
Drug: Pantoprazole — 40 mg x 1 daily intravenously from ICU admission to ICU discharge
  Other Names: Pantoloc
  Arms: Proton pump inhibitor (PPI)
Other: Saline (0.9%) — 10 ml of isotonic saline x 1 daily intravenously from ICU admission to ICU discharge
  Arms: Normal saline

SUMMARY:
Stress ulcer prophylaxis (SUP) is standard of care in the intensive care unit (ICU), however the quantity and quality of evidence is low and potential harm has been reported.

The aim of the SUP-ICU trial is to asses the overall benefits and harms of SUP with proton pump inhibitor in adult critically ill patients in the ICU.

DETAILED DESCRIPTION:
Critically ill patients in the ICU are at risk of stress related gastrointestinal (GI) bleeding, and SUP is recommended. However, the quantity and quality of evidence supporting SUP is low and has been questioned. Furthermore studies have shown that proton pump inhibitors (PPIs) may increase the risk of pneumonia, clostridium difficile infection and acute myocardial ischemia. The aim of the SUP-ICU trial is to assess the benefits and harms of SUP with PPI in adult critically ill patients in the ICU.

ELIGIBILITY:
INCLUSION CRITERIA:

* Acute admission to the ICU
* Age ≥ 18 years
* One or more of the following risk factors:

  * Shock (continuous infusion with vasopressors or inotropes, systolic blood pressure < 90 mmHg, mean arterial blood pressure < 70 mmHg or lactate > 4 mmol/l)
  * Acute or chronic intermittent or continuous renal replacement therapy
  * Invasive mechanical ventilation which is expected to last > 24 hours
  * Coagulopathy (platelets < 50 x 109/l or international normalized ratio (INR) > 1.5 or prothrombin time (PT) > 20 seconds) documented within the last 24 hours
  * Ongoing treatment with anticoagulant drugs (prophylaxis doses excluded)
  * History of coagulopathy (platelets < 50 x 109/l or INR > 1.5 or PT > 20 seconds) within 6 months prior to hospital admission
  * History of chronic liver disease (portal hypertension, cirrhosis proven by biopsy, computed tomography (CT) scan or ultrasound, history of variceal bleeding or hepatic encephalopathy in the past medical history)

EXCLUSION CRITERIA:

* Contraindications to PPI
* Ongoing treatment with PPI and/or H2RA on a daily basis
* GI bleeding of any origin during current hospital admission
* Diagnosed with peptic ulcer during current hospital admission
* Organ transplant during current hospital admission
* Withdrawal from active therapy or brain death
* Fertile woman with positive urine human chorionic gonadotropin (hCG) or plasma-hCG
* Consent according to national regulations not obtainable

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3350 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2017-10-22 (Actual); Study Completion 2018-01-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Morten Hylander Møller, MD, PhD, Principal Investigator — Rigshospitalet, Denmark; Anders Perner, MD, PhD, Study Chair — Rigshospitalet, Denmark
Locations (33):
- Denmark (19):
  - Dept. of Intensive Care, Aalborg University Hospital, Aalborg
  - Dept. of Intensive Care, Århus University Hospital Nørrebrogade, Aarhus
  - Dept. of Intensive Care, Århus University Hospital Skejby, Aarhus
  - Dept. of Intensive Care 4131, Copenhagen University Hospital Rigshospitalet, Copenhagen
  - Dept. of Neurointensive Care, Copenhagen University Hospital Rigshospitalet, Copenhagen
  - Dept. of Intensive Care, Bispebjerg Hospital, Copenhagen
  - Dept. of Intensive Care, Copenhagen University Hospital Herlev, Herlev
  - Dept. of Intensive Care, Herning Hospital, Herning
  - Dept. of Intensive Care, Hillerød Hospital, Hillerød
  - Dept. of Intensive Care, Hjørring Hospital, Hjørring
  - Dept. of Intensive Care, Holbæk Hospital, Holbæk
  - Dept. of Intensive Care, Holstebro Hospital, Holstebro
  - Dept. of Intensive Care, Køge University Hospital, Køge
  - Dept. of Intensive Care, Nykøbing Falster Sygehus, Nykøbing Falster
  - Dept. of Intensive Care, Randers Hospital, Randers
  - Dept. of Intensive Care, Roskilde Hospital, Roskilde
  - Dept. of Intensive Care, Slagelse Hospital, Slagelse
  - Dept. of Intensive Care, Vejle Hospital, Vejle
  - Dept. of Intensive Care, Viborg Hospital, Viborg
- Finland (5):
  - Dept. of Intensive Care, Helsinki University Hospital, Helsinki
  - Dept. of Intensive Care, Kuopio University Hospital, Kuopio
  - Dept. of Intensive Care, Oulu University Hospital, Oulu
  - Dept. of Intensive Care, Tampere University Hospital, Tampere
  - Dept. of Intensive Care, Turku University Hospital, Turku
- Netherlands (2):
  - Dept. of Intensive Care, University Medical Center Groningen, Groningen
  - Dept. of Intensive Care, Heerlen Hospital, Heerlen
- Norway (4):
  - Dept. of Intensive Care, Bergen University Hospital, Bergen
  - Dept. of Intensive Care, Akershus University Hospital, Lørenskog
  - Dept. of Intensive Care, Oslo University Hospital, Oslo
  - Dept. of Intensive Care, Stavanger University Hospital, Stavanger
- Switzerland (2):
  - Dept. of Intensive Care, Basel University Hospital, Basel
  - Dept. of Intensive Care, Bern University Hospital, Bern
- Dept. of Intensive Care, University Hospital of Wales, Cardiff, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Krag M, Perner A, Wetterslev J, Wise MP, Hylander Moller M. Stress ulcer prophylaxis versus placebo or no prophylaxis in critically ill patients. A systematic review of randomised clinical trials with meta-analysis and trial sequential analysis. Intensive Care Med. 2014 Jan;40(1):11-22. doi: 10.1007/s00134-013-3125-3. Epub 2013 Oct 19. PMID 24141808
- [Background] Krag M, Perner A, Wetterslev J, Wise MP, Borthwick M, Bendel S, McArthur C, Cook D, Nielsen N, Pelosi P, Keus F, Guttormsen AB, Moller AD, Moller MH; SUP-ICU co-authors. Prevalence and outcome of gastrointestinal bleeding and use of acid suppressants in acutely ill adult intensive care patients. Intensive Care Med. 2015 May;41(5):833-45. doi: 10.1007/s00134-015-3725-1. Epub 2015 Apr 10. PMID 25860444
- [Derived] Halling CMB, Moller MH, Marker S, Krag M, Kjellberg J, Perner A, Gyrd-Hansen D. The effects of pantoprazole vs. placebo on 1-year outcomes, resource use and employment status in ICU patients at risk for gastrointestinal bleeding: a secondary analysis of the SUP-ICU trial. Intensive Care Med. 2022 Apr;48(4):426-434. doi: 10.1007/s00134-022-06631-2. Epub 2022 Feb 5. PMID 35122105
- [Derived] Granholm A, Marker S, Krag M, Zampieri FG, Thorsen-Meyer HC, Kaas-Hansen BS, van der Horst ICC, Lange T, Wetterslev J, Perner A, Moller MH. Heterogeneity of treatment effect of prophylactic pantoprazole in adult ICU patients: a post hoc analysis of the SUP-ICU trial. Intensive Care Med. 2020 Apr;46(4):717-726. doi: 10.1007/s00134-019-05903-8. Epub 2020 Jan 14. PMID 31938829
- [Derived] Granholm A, Lange T, Anthon CT, Marker S, Krag M, Meyhoff TS, Wise MP, Borthwick M, Bendel S, Keus F, Guttormsen AB, Schefold JC, Wetterslev J, Perner A, Moller MH. Time to onset of gastrointestinal bleeding in the SUP-ICU trial: A pre-planned substudy. Acta Anaesthesiol Scand. 2019 Nov;63(10):1346-1356. doi: 10.1111/aas.13459. Epub 2019 Sep 11. PMID 31441031
- [Derived] Granholm A, Marker S, Krag M, Zampieri FG, Thorsen-Meyer HC, Kaas-Hansen BS, van der Horst ICC, Lange T, Wetterslev J, Perner A, Moller MH. Heterogeneity of treatment effect of stress ulcer prophylaxis in ICU patients: A secondary analysis protocol. Acta Anaesthesiol Scand. 2019 Oct;63(9):1251-1256. doi: 10.1111/aas.13432. Epub 2019 Jul 18. PMID 31321771
- [Derived] Marker S, Krag M, Perner A, Wetterslev J, Lange T, Wise MP, Borthwick M, Bendel S, Keus F, Guttormsen AB, Schefold JC, Rasmussen BS, Elkmann T, Bestle M, Arenkiel B, Laake JH, Kamper MK, Lang M, Pawlowicz-Dworzanska MB, Karlsson S, Liisanantti J, Dey N, Knudsen H, Granholm A, Moller MH; SUP-ICU trial investigators. Pantoprazole in ICU patients at risk for gastrointestinal bleeding-1-year mortality in the SUP-ICU trial. Acta Anaesthesiol Scand. 2019 Oct;63(9):1184-1190. doi: 10.1111/aas.13436. Epub 2019 Jul 19. PMID 31282567
- [Derived] Marker S, Perner A, Wetterslev J, Krag M, Lange T, Wise MP, Borthwick M, Bendel S, Keus F, Guttormsen AB, Schefold JC, Moller MH; SUP-ICU investigators. Pantoprazole prophylaxis in ICU patients with high severity of disease: a post hoc analysis of the placebo-controlled SUP-ICU trial. Intensive Care Med. 2019 May;45(5):609-618. doi: 10.1007/s00134-019-05589-y. Epub 2019 Mar 12. PMID 30863936
- [Derived] Krag M, Marker S, Perner A, Wetterslev J, Wise MP, Schefold JC, Keus F, Guttormsen AB, Bendel S, Borthwick M, Lange T, Rasmussen BS, Siegemund M, Bundgaard H, Elkmann T, Jensen JV, Nielsen RD, Liboriussen L, Bestle MH, Elkjaer JM, Palmqvist DF, Backlund M, Laake JH, Badstolokken PM, Gronlund J, Breum O, Walli A, Winding R, Iversen S, Jarnvig IL, White JO, Brand B, Madsen MB, Quist L, Thornberg KJ, Moller A, Wiis J, Granholm A, Anthon CT, Meyhoff TS, Hjortrup PB, Aagaard SR, Andreasen JB, Sorensen CA, Haure P, Hauge J, Hollinger A, Scheuzger J, Tuchscherer D, Vuilliomenet T, Takala J, Jakob SM, Vang ML, Paelestik KB, Andersen KLD, van der Horst ICC, Dieperink W, Fjolner J, Kjer CKW, Solling C, Solling CG, Karttunen J, Morgan MPG, Sjobo B, Engstrom J, Agerholm-Larsen B, Moller MH; SUP-ICU trial group. Pantoprazole in Patients at Risk for Gastrointestinal Bleeding in the ICU. N Engl J Med. 2018 Dec 6;379(23):2199-2208. doi: 10.1056/NEJMoa1714919. Epub 2018 Oct 24. PMID 30354950
- [Derived] Krag M, Perner A, Wetterslev J, Wise MP, Borthwick M, Bendel S, Pelosi P, Keus F, Guttormsen AB, Schefold JC, Moller MH; SUP-ICU investigators. Stress ulcer prophylaxis with a proton pump inhibitor versus placebo in critically ill patients (SUP-ICU trial): study protocol for a randomised controlled trial. Trials. 2016 Apr 19;17(1):205. doi: 10.1186/s13063-016-1331-3. PMID 27093939

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Proton Pump Inhibitor (PPI) | Normal Saline
Started (52 patients were randomised in error BEFORE receiving the first dose of IMP/placebo. 3350-52=3298) | 1645 | 1653
Completed (1644/1647 in the secondary outcome analyses 1642/1640 in the primary outcome analysis) | 1644 | 1647
Not Completed | 1 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Proton Pump Inhibitor (PPI) | Normal Saline | Total
Number analyzed (Participants) | 1644 | 1647 | 3291
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 67 [56 to 75] | 67 [55 to 75] | 67 [55 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 605 | 580 | 1185
  Male | 1039 | 1067 | 2106
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1644 | 1647 | 3291
Region of Enrollment [Number; unit: participants]
  Netherlands | 88 | 84 | 172
  Norway | 96 | 101 | 197
  Finland | 128 | 130 | 258
  Denmark | 1061 | 1064 | 2125
  United Kingdom | 34 | 33 | 67
  Switzerland | 237 | 235 | 472

OUTCOME MEASURES:

1. Primary Outcome: Mortality
Description: Landmark mortality 90-days after randomization
Time Frame: 90 days
Population: Intention-to-treat
Measure: Count of Participants; unit: Participants
Arm/Group | Proton Pump Inhibitor (PPI) | Normal Saline
Number analyzed (Participants) | 1642 | 1640
Participants | 510 | 499

2. Secondary Outcome: Number of Participants With Clinically Important GI Bleeding, Pneumonia, Clostridium Difficile Infection or Acute Myocardial Ischemia
Description: Composite outcome of the number of participants with one or more of the mentioned conditions in the ICU
Time Frame: Until ICU discharge, maximum 90 days
Population: Intention-to-treat
Measure: Count of Participants; unit: Participants
Arm/Group | Proton Pump Inhibitor (PPI) | Normal Saline
Number analyzed (Participants) | 1644 | 1647
Participants | 360 | 372

3. Secondary Outcome: Number of Participants With Clinically Important GI Bleeding
Description: Number of participants with one or more episodes of clinically important GI bleeding in the ICU
Time Frame: Until ICU discharge, maximum 90 days
Measure: Count of Participants; unit: Participants
Arm/Group | Proton Pump Inhibitor (PPI) | Normal Saline
Number analyzed (Participants) | 1644 | 1647
Participants | 41 | 69

4. Secondary Outcome: Number of Participants With One or More Infectious Adverse Events
Description: Number of participants with one or more episodes of pneumonia or clostridium difficile infection in the ICU
Time Frame: Until ICU discharge, maximum 90 days
Measure: Count of Participants; unit: Participants
Arm/Group | Proton Pump Inhibitor (PPI) | Normal Saline
Number analyzed (Participants) | 1644 | 1647
Participants | 276 | 279

5. Secondary Outcome: Mortality
Description: Data for landmark mortality 1 year after randomization.
Time Frame: 1 year
Population: Twenty-one patients were lost to follow-up, as compared to the primary outcome (90-day mortality): 7 patients in the PPI arm and 14 patients in the placebo arm
Measure: Count of Participants; unit: Participants
Arm/Group | Proton Pump Inhibitor (PPI) | Normal Saline
Number analyzed (Participants) | 1635 | 1626
Participants | 610 | 601

6. Secondary Outcome: Percentage of Days Alive Without Organ Support
Description: Percentage of days alive and free from mechanical ventilation, circulatory support and renal replacement therapy
Time Frame: Within 90 days
Measure: Number; unit: percentage of days
Arm/Group | Proton Pump Inhibitor (PPI) | Normal Saline
Number analyzed (Participants) | 1644 | 1647
percentage of days | 92 | 92

7. Secondary Outcome: Number of Serious Adverse Reactions
Description: Serious adverse reactions are: anaphylactic reactions, agranulocytosis, pancytopenia, acute hepatic failure, Steven Johnsons Syndrome and toxic epidermal necrolysis, interstitial nephritis and angioedema.
Time Frame: Until ICU discharge, maximum 90 days
Measure: Count of Participants; unit: Participants
Arm/Group | Proton Pump Inhibitor (PPI) | Normal Saline
Number analyzed (Participants) | 1644 | 1647
Participants | 0 | 0

8. Secondary Outcome: A Health Economic Analysis
Description: This has not been completed yet.
Time Frame: 90 days
Reporting Status: Not Posted, anticipated posting 2025-01

ADVERSE EVENTS:
Time Frame: 90 days (for mortality 1 year)
Arm/Group | Proton Pump Inhibitor (PPI) | Normal Saline
All-Cause Mortality (participants affected / at risk) | 610/1635 | 601/1626
Serious Adverse Events (participants affected / at risk) | 0/1644 | 0/1647
Other Adverse Events (participants affected / at risk) | 360/1644 | 372/1647
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Proton Pump Inhibitor (PPI) (N=1644) | Normal Saline (N=1647)
Clinically important events (General disorders) | 360 | 372

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-08-01): https://cdn.clinicaltrials.gov/large-docs/21/NCT02467621/Prot_SAP_000.pdf